CLINICAL TRIAL: NCT02772900
Title: Effect of a Beetroot-based Nutritional Gel on Vascular Function and Forearm Muscle Oxygenation Responses in the Elderly at Cardiometabolic Risk
Brief Title: Aging, Nitrate, Endothelial Function and Muscle Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Thiago Alvares, D.Sc., Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 15510313.5.0000.5257
Record Dates: First submitted 2016-05-02; First posted 2016-05-16 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Aging; Hypertension; Dyslipidemia; Abdominal Obesity
Keywords: Aging; Beetroot; Dietary Nitrate; Functional Food; Vascular Function
MeSH Terms: conditions — Hypertension; Dyslipidemias; Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Beetroot gel (dietary nitrate) (Active Comparator): Beetroot-based nutritional gel containing approximately 10.0 mmol of nitrate per dose
  Interventions: Other: Beetroot-based nutritional gel
- Placebo gel (nitrate-depleted) (Active Comparator): Nutritional gel nitrate-depleted
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Beetroot-based nutritional gel — 100 g of beetroot-based nutritional gel containing approximately 12 mmol of nitrate.
  Arms: Beetroot gel (dietary nitrate)
Other: Placebo — 100 g of apple-based nutritional gel containing approximately 0.02 mmol of nitrate.
  Arms: Placebo gel (nitrate-depleted)

SUMMARY:
Aging has been associated with reduced bioavailability of nitric oxide (NO) and endothelial dysfunction. Beetroot consumption, a nitrate-rich food, has been associated with increased NO bioconversion, which may promote beneficial effects on vascular health. The present study evaluated the effects of a beetroot-based nutritional gel (BG) on vascular function, arterial stiffness and blood pressure in the elderly at cardiometabolic risk. Twenty elderly individuals were submitted to BG and nitrate-depleted gel (PLA) interventions. Brachial flow-mediated dilation (FMD), blood flow velocity (BFV), peak wave velocity (PWVβ), augmentation index (AI), stiffness parameter (β), pressure-strain elasticity modulus (Ep), arterial compliance (AC), muscle oxygenation and function were measured 90 min after interventions. Urinary nitrate, nitrite, systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) were measured at baseline, 90 min and 150 min after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Elderly participants (≥ 65 years)
* Taking between 1 and 3 anti-hypertensive medications for high blood pressure;
* Elevated triglycerides ≥ 150 mg/dL;
* Reduced HDL-cholesterol < 50 mg/dL for women and < 40 mg/dL for men;
* Elevated waist circumference by population definition (male: > 102 cm and female: > 88 cm).

Exclusion Criteria: elevated fasting glucose (≥ 100 mg/dL), smoking, beetroot allergy, unwillingness to avoid beetroot products during the entire study, other chronic diseases (diabetes, liver disease, etc.), or acutely ill.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in endothelial function as evaluated by the flow-mediated dilation. | Evaluated 120 min after the nutritional intervention
Changes in the arterial stiffness as evaluated by the peak wave velocity. | Evaluated 120 min after the nutritional intervention
Changes in the clinical blood pressure | Evaluated before, 120 min and 180 min after the nutritional intervention
Changes in the muscle oxygenation as evaluated by the levels of oxygenated | Evaluated 150 min after the nutritional intervention
Changes in the muscle function as evaluated by the maximal voluntary contraction of the forearm muscle | Evaluated before and 180 min after the nutritional intervention
Changes in endothelial function as evaluated by blood flow velocity | Evaluated 120 min after the nutritional intervention
Changes in endothelial function as evaluated by reactive hyperemia. | Evaluated 120 min after the nutritional intervention
Changes in the arterial stiffness as evaluated by augmentation index | Evaluated 120 min after the nutritional intervention
Changes in the arterial stiffness as evaluated by the stiffness parameter | Evaluated 120 min after the nutritional intervention
Changes in the arterial stiffness as evaluated by the pressure-strain elasticity modulus | Evaluated 120 min after the nutritional intervention
Changes in the arterial stiffness as evaluated by the arterial compliance. | Evaluated 120 min after the nutritional intervention
Changes in the muscle oxygenation as evaluated by the levels of deoxygenated hemoglobin | Evaluated 150 min after the nutritional intervention